CLINICAL TRIAL: NCT00493428
Title: Treatment of Non-Metastatic Hepatocellular Carcinoma in Humans by Increasing Gabaergic Activity: A Pilot Study
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study have been stoped because the protocol is going to be modify.
Sponsor: University of Manitoba (Other)
Responsible Party: Minuk Gerald, Liver Unit, Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2006:156
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; GABAergic Activity; Baclofen
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Baclofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Baclofen — Patients will receive an initial dose of: 5 mg tid to be increased as tolerated to a maximum dose of 20 mg qid. This dose range and schedule reflects that suggested for the drug's muscle relaxant properties in human.
  Other Names: Lioresal,Nu-Baclo

SUMMARY:
Recent studies indicate that liver cancer cells possess a receptor called the GABA-B receptor that when activated, inhibits the spread of cancer cells in test tubes. One of the drugs that activate these receptors is Baclofen, an agent that was originally developed to treat patients with various neurologic disorders. In this study, patients with recently identified liver cancer will be treated with Baclofen in an attempt to prevent or delay spread of the cancer beyond the liver. The time it takes for liver cancer to spread in the patients will be compared to the results obtained from patients enrolled in previous studies where Baclofen was not used.

DETAILED DESCRIPTION:
A total of 47 consecutive patients with radiologic or histologic evidence of non metastatic liver cancer will be enrolled over a 2-4 year period. Subjects will receive oral Baclofen at the manufacturer's suggested maximal dose. Clinical, hematologic, biochemical, and radiologic features of liver function, tumor metastasis and recurrence will be monitored at regular time intervals over a 2 year treatment period. The primary study end point will be the event of interest (time to metastasis or recurrence). Secondary end points will include time to metastasis following recurrence, objective tumor responses (complete, partial and non response), response duration, survival and safety. It is hoped the results of this study will permit liver cancer patients to remain candidates for surgical resection and transplantation longer than would otherwise have been the case.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of HCC and no evidence of extra-hepatic metastases on CT/MRI scan of the abdomen, CT of the chest and brain and a negative bone scan.
* Patients undergoing local therapy (resection, ablation or chemoembolization) and those listed for liver transplantation will not be excluded from participating in the study.
* Patients with multiple space occupying lesions within the liver (but no evidence of extra-hepatic metastases) will continue to be eligible (the distinction between regenerative nodules and multi-focal HCC versus intra-hepatic metastases can not be made with certainty by presently available techniques).
* Karnofsky Performance Status (KPS) ≥ 60 %.
* Age 18 years or greater.
* Life expectancy of at least 12 weeks.
* Concomitant Medications
* Patients should be on stable doses of other medications (no change in dose for two weeks prior to study initiation) when entered into the study.
* Patient consent must be obtained from all patients prior to entry into the trial.
* Patients must be accessible for treatment and follow-up i.e. residing within reasonable geographical limits of the study site.

Exclusion Criteria:

* Any investigational agent within a minimum of 6 weeks prior to study treatment.
* Pregnant or lactating women; women or men of childbearing potential unless using effective contraception. Patients capable of reproduction must agree to use appropriate methods of contraception during the study and for six months afterwards. Female patients of childbearing potential must have a negative urine pregnancy test within 14 days of study enrollment.
* Patients whose partners are pregnant.
* Other serious illness or medical conditions which would not permit the patient to be managed according to the protocol including:

  * History of a psychiatric disorder which would impair the ability to obtain consent or follow-up tumor imaging.
  * Active uncontrolled infection.
* Any known defect in GABA metabolism or hypersensitivity to Baclofen.
* Patients with previous organ allograft or taking immunomodulatory drugs.
* Renal failure not being managed by dialysis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Document and Compare the effects of the GABAb receptor agonist Baclofen on the time to develop tumor metastasis in patients with non-metastatic HCC at diagnosis who subsequently undergo surgical resection, ablation or chemoembolization. | 6 years

SECONDARY OUTCOMES:
Document and compare the effects of the GABAb receptor agonist Baclofen on changes in serum tumor markers ( alpha-fetoprotein andd CA19-9 levels) in patients with no-metastatic HCC at diagnosis. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Minuk Y Minuk, MD, FRCPC, Principal Investigator — University of Manitoba
Locations (2):
- Canada (2):
  - Liver Unit, Section of Hepatology, Department of Medicine,Health Sciences Centre, Winnipeg, Manitoba
  - Liver Unit, health sciences Centre, Winnipeg, Manitoba